CLINICAL TRIAL: NCT07060469
Title: Comparative Analysis of Anatomic Shoulder Arthroplasty, Hemiarthroplasty, and Reverse Shoulder Arthroplasty in Patients Over 70: A Retrospective Single Unit Single Surgeon Study
Brief Title: Comparison Between Anatomic Shoulder Arthroplasty, Hemiarthroplasty, and Reverse Shoulder Arthroplasty.
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 905; RL1 905 (Other: The Robert Jones and Agnes Hunt Orthopaedic Hospital)
Record Dates: First submitted 2025-04-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anatomic Shoulder Arthroplasty: Type of shoulder replacement
- Hemiarthroplasty: Type of shoulder replacement
- Reverse Shoulder Arthroplasty: Type of shoulder replacement

SUMMARY:
This study aims to evaluate outcomes in patients over 70 years of age who underwent anatomic shoulder arthroplasty, hemiarthroplasty, or reverse shoulder arthroplasty, focusing on revision rates, rotator cuff integrity as primary and Oxford Shoulder Scores as secondary outcome measures.

DETAILED DESCRIPTION:
Despite numerous studies, the literature presents conflicting evidence regarding the comparative effectiveness of anatomic shoulder arthroplasty (aTSA) versus reverse shoulder arthroplasty in primary humeral osteoarthritis among patients aged over 70 years.

There is anecdotal evidence that doing a shoulder replacement in the above 70-year-old patient could potentially lead to early failure and revision due to rotator cuff tears. There is currently a UK run RCT looking into randomising patient above 60 in reverse or anatomic shoulder replacement. Current literature provides inconclusive evidence, and our local practice does not suggest early failure and revision of anatomic shoulder replacement in the over 70s. The aim of the study is to investigate this and provide solid evidence.

This retrospective analysis will utilize a decade of data from a single surgeon's practice, supplemented by information retrieved from the UK National Joint Registry in. Patients that had a shoulder replacement-anatomic, reverse, or hemi-arthroplasty-aged over 70 at the time of surgery will be included. Data will be cross-referenced with local databases for pre- and postoperative Oxford Shoulder Scores (OSS), primary diagnoses, and complications. The study population includes patients with recorded Oxford Shoulder Scores at a minimum of one year and a maximum of seven years postoperatively. IBM SPSS V.25 will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

All genders Over 70 All ethnic groups Anatomic / Reverse / Hemi shoulder replacement

Exclusion Criteria:

Under 70 years of age Shoulder replacement for trauma/tumour

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients who have had a shoulder replacement within the last 10 years anatomic, reverse, or hemi-arthroplasty and who are aged over 70 at the time of surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff failure | within the last 10 years
  Information will be retrieved from the UK National Joint Registry in. Patients that had a shoulder replacement-anatomic, reverse, or hemi-arthroplasty. This will indicate the failure rate of these types of shoulder replacement.

SECONDARY OUTCOMES:
Oxford Shoulder Score (OSS) | within the last 7 years
  The study population includes patients with recorded Oxford Shoulder Scores at a minimum of one year and a maximum of seven years postoperatively. The lower the score indicates the greatest disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mr I Tsolis, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao KA, Boschert EN, O'Keefe DS, Saengchote SA, Schoch BS, Wright JO, Wright TW, Farmer KW, Struk AM, King JJ. Comparison of clinical outcomes of revision reverse total shoulder arthroplasty for failed primary anatomic vs. reverse shoulder arthroplasty. JSES Int. 2022 Dec 16;7(2):257-263. doi: 10.1016/j.jseint.2022.11.003. eCollection 2023 Mar. PMID 36911771
- [Background] Heifner JJ, Kumar AD, Wagner ER. Glenohumeral osteoarthritis with intact rotator cuff treated with reverse shoulder arthroplasty: a systematic review. J Shoulder Elbow Surg. 2021 Dec;30(12):2895-2903. doi: 10.1016/j.jse.2021.06.010. Epub 2021 Jul 20. PMID 34293419
- [Background] Orvets ND, Chan PH, Taylor JM, Prentice HA, Navarro RA, Garcia IA. Similar rates of revision surgery following primary anatomic compared with reverse shoulder arthroplasty in patients aged 70 years or older with glenohumeral osteoarthritis: a cohort study of 3791 patients. J Shoulder Elbow Surg. 2023 Sep;32(9):1893-1900. doi: 10.1016/j.jse.2023.03.021. Epub 2023 Apr 17. PMID 37075936
- [Background] Su F, Nuthalapati P, Feeley BT, Lansdown DA. Outcomes of anatomic and reverse total shoulder arthroplasty in patients over the age of 70: a systematic review. JSES Rev Rep Tech. 2023 Mar 4;3(2):181-188. doi: 10.1016/j.xrrt.2023.02.003. eCollection 2023 May. PMID 37588441
- [Background] Jensen AR, Tangtiphaiboontana J, Marigi E, Mallett KE, Sperling JW, Sanchez-Sotelo J. Anatomic total shoulder arthroplasty for primary glenohumeral osteoarthritis is associated with excellent outcomes and low revision rates in the elderly. J Shoulder Elbow Surg. 2021 Jul;30(7S):S131-S139. doi: 10.1016/j.jse.2020.11.030. Epub 2021 Jan 20. PMID 33484829